CLINICAL TRIAL: NCT05294822
Title: Autologous Regenerative Islet Transplantation for Insulin-dependent Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZXHZ-IIT-01
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous regenerative islet transplantation for insulin-dependent diabetes mellitus (Experimental)
  Interventions: Procedure: Autologous regenerative islet transplantation for insulin-dependent diabetes mellitus

INTERVENTIONS:
Procedure: Autologous regenerative islet transplantation for insulin-dependent diabetes mellitus — Islet transplantation was completed using percutaneous transhepatic portal vein puncture. After transplantation, rabbit anti human thymocyte immunoglobulin (ATG) or basiliximab was used as induction therapy and low-dose tacrolimus combined with sirolimus or mycophenolate mofetil were used as immunosuppressive maintenance therapy.

SUMMARY:
This is a single-center, phase IIT clinical trial to evaluate autologous regenerative islet transplantation for insulin-dependent diabetes mellitus.

Twenty patients with insulin-dependent diabetes mellitus will be enrolled: poor blood glucose control despite intensive exogenous insulin therapy. The primary endpoint will be defined by the return to normal blood glucose control without insulin at 12 months after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Insulin-dependent diabetes mellitus, the specific criteria are (1 of 4-6 is sufficient).

  1. Age: 18-70 years old;
  2. History of diabetes mellitus >1 year;
  3. Insulin-dependent and total daily insulin dose >20 units;
  4. Poor blood glucose control despite intensive exogenous insulin therapy (or high blood glucose fluctuation, glycation >8% );
  5. Frequent hypoglycemic episodes with unconsciousness; 6) Diabetic nephropathy, patients who need to receive kidney transplantation.

Exclusion Criteria:

* 1) Severe heart disease; 2) Severe mental disorders, poor compliance or alcohol abuse; 3) Active infection or with malignancy; 4) Weight greater than 25% of ideal weight; 5) Evidence of endogenous insulin secretion, such as type 2 diabetes; 6) Smoking; 7) During gestation or preparation for gestation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in C-peptide | before surgery, once a week for the first month after surgery, once a month between the second and six month after surgery, and once every 3 months afterwards, with the follow-up time of 12 months in total
  Changes in C-peptide (fasting C-peptide and post-stimulated C-peptide) of patients during the study period since baseline.
Changes in insulin | before surgery, once a week for the first month after surgery, once a month between the second and six month after surgery, and once every 3 months afterwards, with the follow-up time of 12 months in total
  Changes in insulin (fasting insulin and post-stimulated insulin) of patients during the study period since baseline.
Changes in HbA1c values | before surgery, once a week for the first month after surgery, once a month between the second and six month after surgery, and once every 3 months afterwards, with the follow-up time of 12 months in total
  Changes in HbA1c values of patients during the study period since baseline.

SECONDARY OUTCOMES:
Change in the patient's daily insulin unit requirement | Data will be recorded every day after the surgery until insulin treatment stops during the follow-up time of 12 months.
  Change in the patient's daily insulin unit requirement during the study period.
Number of severe hypoglycemic events | Data will be recorded every week after the surgery during the follow-up time of 12 months.
  Number of severe hypoglycemic events in patients during the study period.
Changes in glucagon | before surgery, once a week for the first month after surgery, once a month between the second and six month after surgery, and once every 3 months afterwards, with the follow-up time of 12 months in total
  Changes in glucagon since baseline during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yin, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided